CLINICAL TRIAL: NCT02863159
Title: A Clinical Assessment of the Full Range of Functional Vision (Distance, Intermediate, Near) With Three Tecnis Multifocal IOL 1-Piece Models [+2.75D (ZKB00), +3.25D (ZLB00), +4.00D (ZMB00)] in Subjects Undergoing Bilateral Cataract Extraction
Brief Title: A Clinical Assessment of the Full Range of Functional Vision With Three Tecnis Multifocal IOL 1-Piece Models in Bilateral Cataract Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dell Laser Consultants (Other)
Collaborators: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SJDLA-2015-01
Record Dates: First submitted 2016-03-08; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Active Comparator): 50 qualified study patients will receive the +2.75D (ZKB00) in their dominant eye and the +3.25D (ZLB00) in their non-dominant eye.
  Interventions: Device: Tecnis Multifocal 1-Piece IOL
- Treatment Group 2 (Active Comparator): 50 qualified study patients will receive the +2.75D (ZKB00) in their dominant eye and the +4.00D (ZMB00) in their non-dominant eye.
  Interventions: Device: Tecnis Multifocal 1-Piece IOL

INTERVENTIONS:
Device: Tecnis Multifocal 1-Piece IOL — +2.75D (ZKB00), +3.25D (ZKB00), +4.00D (ZMB00)

SUMMARY:
The objective of this study is to evaluate the uncorrected binocular distance, intermediate, and near visual acuities, and assess patient's spectacle independence and satisfaction in individuals undergoing bilateral cataract extraction that have received two different arms of near add design IOLs of the same diffractive multifocal model.

DETAILED DESCRIPTION:
This will be a multi-center, parallel comparison clinical study design with two treatment groups. One hundred (100) qualified study patients will receive a +2.75D (ZKB00) Tecnis Multifocal 1-Piece IOL in their dominant eye. Of these study patients, 50 patients will receive the +3.25D (ZLB00) Tecnis Multifocal 1-Piece IOL in their non-dominant eye and the other 50 patients will receive the +4.00D (ZMB00) Tecnis Multifocal 1-Piece IOL in their non-dominant eye. each study patient will undergo the same routine cataract extraction procedures for each eye, with the second eye scheduled to undergo cataract extraction within 7 to 30 days after the first eye. In addition, as is customary for the surgeon, each study patient will receive the same open-label pre-operative, operative and post-operative medications over the course of the study period.

ELIGIBILITY:
Inclusion Criteria:

* A patient with bilateral cataracts for which phacoemulsification extraction and a posterior multifocal IOL implantation has been planned for both eyes.
* Male or female in good general health, 21 years of age or older at the time of the pre-operative examination and willing to have surgery on their second eye within 7 to 30 days of their first eye.
* A patient must be willing to comply with study instructions, agree to make all office appointments, and complete the entire course of the study.
* A patient has the visual potential of 20/32 or better in each eye after cataract removal and IOL implantation in the judgment of the investigator.
* A patient with a preoperative corneal astigmatism of ≤ 1.5D in each eye [intraoperative management of corneal astigmatism is permissible, and may include arcuate incision(s) or LRI(s).]
* A patient has a post-operative astigmatism target of ≤ 0.5D in each eye.
* A patient with clear ocular media other than cataract in each eye.
* A patient with normal OCT of the macula in each eye or a macula judged to be normal by the investigator by clinical examination.
* A patient with naturally dilated pupil sizes of > 3.5mm, evaluated under mesopic illumination.
* A patient must be able to read, comprehend and be willing to give HIPAA and Informed Consent.

Exclusion Criteria:

* A patient with a known pathology that may affect visual acuity (as determined by the investigator); particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.) in either eye.
* A patient with amblyopia or strabismus.
* A patient with capsular or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome) in either eye.
* A patient with pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate as least 3.5mm under mesopic/scotopic conditions) in either eye.
* A patient with evidence of Epithelial Basement Membrane Dystrophy on slit-lamp examination in either eye.
* A patient with evidence of keratoconus or significant irregular astigmatism on pre-operative topography in either eye.
* A patient with a history of ocular trauma, or ocular surgery in either eye.
* A patient that may, or is expected to undergo surgical intervention and/or ocular laser treatment prior to or during the study period in either eye.
* A patient that had refractive surgery (LASIK, LASEK, RK, PRK, etc.) prior to cataract surgery in either eye.
* A patient with a history of wearing PMMA lenses within 6 months, gas permeable lenses within one month, or extended wear daily soft contact lenses within seven days of their scheduled surgery.
* A patient that requires the use of systemic or ocular medications that may affect vision.
* A patient with an uncontrolled acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes, immunocompromised, etc.).
* A patient with any uncontrolled systemic disease. A potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
* A patient currently participating or who has participated within 30 days prior to the start of this study in a drug or other investigational research study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Measurements of uncorrected and best corrected visual acuities under mesopic illumination at distance, intermediate, and near using the ETDRS chart. | 90 days post-operative
  Uncorrected visual acuity measured under mesopic illumination using the ETDRS chart at 4 meters, 66.7cm, and 40.0 cm. Best-corrected visual acuity measured under mesopic illumination using the ETDRS chart at 4 meters, 66.7 cm, and 40.0 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Dell, MD, Principal Investigator — Dell Laser Consultants
Locations (1):
- Dell Laser Consultants, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dell SJ. Evaluation of Visual and Subjective Outcomes with Mix-and-Match of Three One-Piece Tecnis Multifocal IOLs of Varying Add Powers. Clin Ophthalmol. 2020 Sep 29;14:2903-2911. doi: 10.2147/OPTH.S266120. eCollection 2020. PMID 33061276